CLINICAL TRIAL: NCT06543966
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Phase III Study to Evaluate the Efficacy and Safety of Aprepitant Injection in the Prevention of Post-operative Nausea and Vomiting
Brief Title: Efficacy and Safety Study of Aprepitant Injection for Prevention of Post-operative Nausea and Vomiting
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYH9053-002
Record Dates: First submitted 2024-07-17; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Post-operative Nausea and Vomiting (PONV)
MeSH Terms: conditions — Vomiting | interventions — Aprepitant

STUDY DESIGN:
Intervention Model Description: Parrallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aprepitant Injection (Experimental): Before anesthesia induction, 4.4ml(32mg） was given by a single intravenous injection, which was completed within 30 seconds
  Interventions: Drug: Aprepitant Injection
- Placebo (Placebo Comparator): Before anesthesia induction, 4.4ml(0mg）was given by a single intravenous injection, which was completed within 30 seconds
  Interventions: Drug: Aprepitant Injection Placebo

INTERVENTIONS:
Drug: Aprepitant Injection — Before anesthesia induction, 4.4ml(32mg） was given by a single intravenous injection, which was completed within 30 seconds
  Arms: Aprepitant Injection
Drug: Aprepitant Injection Placebo — Before anesthesia induction, 4.4ml(0mg） was given by a single intravenous injection, which was completed within 30 seconds
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, multi-center phase III study to compare the efficacy and safety of aprepitant injection and placebo in the prevention of post-operative nausea and vomiting (PONV).,

DETAILED DESCRIPTION:
In this study, a randomized, double-blind, placebo-controlled multicenter study will be conducted to evaluate the efficacy and safety of aprepitant injection in the prevention of post-operative nausea and vomiting (PONV).

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 and ≤75 years old; 18 < BMI≤30kg/m^2, body weight ≥45kg; laparoscopic gynecologic or abdominal surgery under general anesthesia that was expected to last at least 1 hour.

expected or agreed to stay in the hospital for 24 hours or more after surgery;

Exclusion Criteria:

diagnostic surgery; scheduled for postoperative transfer to an intensive care unit; requiring placement of a nasogastric or orogastric tube after surgery; Post-operative vomiting may pose significant risk;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Estimated)
Dates: Start 2024-10-28 (Estimated); Primary Completion 2026-03-28 (Estimated); Study Completion 2026-03-28 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rates over 24 hours after the end of surgery | 0-24 hours after the end of surgery
  Complete response (defined as no emetic episodes and no use of rescue therapy)

SECONDARY OUTCOMES:
Proportion of participants who have no nausea in the 0 to 24 hours following the end of surgery | 0-24 hours after the end of surgery
  No nausea（defined as a visual analogue scale (VAS) nausea score < 1.）
Proportion of participants who have significant nausea in the 0 to 24 hours following the end of surgery | 0-24 hours after the end of surgery
  Significant nausea（defined as a visual analogue scale (VAS) nausea score≥4）
Proportion of participants who have no vomiting or retching in the 0 to 24 hours following the end of surgery | 0-24 hours after the end of surgery
  No vomiting or retching（Defined as whether or not use remedy treatment had no vomiting）
Proportion of participants who use the remedial treatment in the 0 to 24 hours following the end of surgery | 0-24 hours after the end of surgery
Time to treatment failure in the 0 to 24 hours following the end of surgery | 0-24 hours after the end of surgery
  defined as the time to the first episode of vomiting (vomiting or retching) or the time to rescue therapy, whichever occurred first.
Proportion of participants who have no vomiting or retching in the 0 to 48 hours following the end of surgery | 0-48 hours after the end of surgery
  No vomiting or retching（Defined as whether or not use remedy treatment had no vomiting）
The time to the first episode of vomiting (vomiting or retching) in the 0 to 48 hours following the end of surgery | 0-48 hours after the end of surgery

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by NIH | Day 0 to Day14
  Safety was assessed by Adverse events (AEs) were recorded after administration.